CLINICAL TRIAL: NCT03156153
Title: A Study of Bumetanide for the Treatment of Children With Autism Spectrum Disorder：a Randomized Double-blind Placebo-controlled Trial
Brief Title: A Study of Bumetanide for the Treatment of Autism Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-16-048
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2019-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Bumetanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bumetanide group (Experimental): Double-blind phase: in the first 3 months, patients will receive the experimental treatment - bumetanide, oral intake, 0.5mg/time, twice a day; Open-label phase: after 3 month double-blined treatment, all the patients will receive 3-month bumetanide treatment - oral intake, 0.5mg/time, twice a day.
  Interventions: Drug: Bumetanide
- Control group (Placebo Comparator): Double-blind phase: in the first 3 months, patients will receive the placebo - oral intake, 0.5mg/time, twice a day; Open-label phase: after 3 month double-blined treatment, patients in this group will receive 3-month bumetanide treatment - oral intake, 0.5mg/time, twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bumetanide — bumetanide tablets, oral intake, 0.5mg, twice daily, respectively at 8 am and 4 pm
  Arms: Bumetanide group
Drug: Placebo — placebo tablets, oral intake, 0.5mg, twice daily, respectively at 8 am and 4 pm
  Arms: Control group

SUMMARY:
The investigators are going to carry out a randomized double-blind placebo-controlled trial to study the efficiency and mechanism of bumetanide on the treatment of children with Autism Spectrum Disorder.

DETAILED DESCRIPTION:
In consideration of the increasing number of autistic children and poor intervention effect in China, it is an urgent to find some effective medicine. Some studies have reported bumetanide, a classic diuretic, could improve autistic behaviors in both animal model and humans; while the efficiency of bumetanide on Chinese autistic chilren is unkonwn and the underlying mechanisms remain unfolding. The investigators aim at investigating whether bumetanide would improve the clinical symptoms in Chinese children with autism within a safe dosage and further study the physiological mechanism beneath.The investigators will regularly assess the participants' autism-related symptoms during medication, as well as the adverse effects of each patient. The investigators will carry out genome-wide association analysis (GWAS) from blood sample, related metabolites in nervous system and compare the concentration of the neurotransmitter in autistic brain before and after 3 months' treatmeat,and also will collect the EEG signal in autistic chilldren when the participants performing certain tasks before and after 3 months' treatment.

ELIGIBILITY:
Inclusion Criteria:

The patients, aged from 3 to 6 years old, were given the diagnosis of ASD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) , by a team of autism experts; Scores for Children Autism Rating Scale (CARS) were more than 30; Signed Informed Consents were provided by parents.

Exclusion Criteria:

Liver and kidney dysfunction; With a history of allergy to sulfa drugs; abnormal ECG; chromosomal abnormality; suffering from nervous system diseases (such as epilepsy, schizophrenia, and so on); using the melatonin treatment for sleep disorders or withdrawal less than three weeks.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale(CARS) | Day 0 and Day 90
  CARS is a behaviour-rating scale used to assess the presence and severity of the symptoms of autism spectrum disorder

SECONDARY OUTCOMES:
Clinical Global Impressions Scale (CGI) | Day 0 and Day 90
  CGI is a scale used to assess the severity of the illness and the global improvement of the patient under intervention
Social Responsiveness Scale (SRS) | Day 0 and Day 90
  SRS is a questionnaire used to assess the presence and severity of social impairment.
Autism Diagnostic Observation Schedule (ADOS) | Day 0 and Day 90
  The ADOS is a structured play session conducted by clinicians, with the total score combines the Social and Communication domain items.
Short Sensory Profile Report | Day 0 and Day 90
  The Sensory Profile is a measure of children's responses to sensory events in daily life. The caregiver completes the Sensory Profile by assessing the frequency of the child's responses to certain sensory processing, modulation, and behavioral/emotional events as described in the 125 items.
Symbolic Play Test | Day 0 and Day 90
  Symbolic Play Test is a nonverbal measure of symbolic functioning in participants aged 12-36 months. The test does not require any expressive speech, and is therefore appropriate for use with all participants with ASD. Participants are sequentially presented with four sets of toys, and their spontaneous manipulation of the objects is observed and recorded on a standardized checklist.
Chinese Communicative Development Inventory | Day 0 and Day 90
  The Chinese Communicative Development Inventories (CCDI) is a questionnaire that is used to direct measures of the participants' language.Change between day 0 and day 90 of the result of the Chinese Communicative Development Inventory

OTHER OUTCOMES:
MRI Structure Imaging and Spectrum imaging, data analysis | Day 0 and Day 90
  Change of structure of the brain and the GABA-neurotransmitters in specific brain regions of the brain.
Multichannel EEG Signals | Day 0 and Day 90
  Change in brain Multichannel EEG signals
Genome wide association study from blood sample | Day 90
  Selection and study of susceptible genes
Analysis of metabolites from blood sample | Day 0 and Day 90
  Metabonomics research

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, doctor, Principal Investigator — Xinhua hospital Affilated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided